CLINICAL TRIAL: NCT06250998
Title: Prediction of Abdominal Aortic Aneurysm Shrinkage After Endovascular Repair With Artificial Intelligence
Brief Title: Prediction of Abdominal Aortic Aneurysm Shrinkage After Stent-placement With Artificial Intelligence
Acronym: ARTinEVAR
Status: Recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: University Medical Center Groningen (Other); Amsterdam UMC, location VUmc (Other); Medisch Spectrum Twente (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1986
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: AAA - Abdominal Aortic Aneurysm
Keywords: AAA; aneurysm shrinkage; EVAR; aneurysm remodeling; artificial intelligence; AI
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to find out what factors contribute to a good treatment outcome in patients who have received a stent for their dilation of the main abdominal artery (abdominal aortic aneurysm or AAA). The primary goal of this study is to build a prediction model for abdominal aortic aneurysm shrinkage one year after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Elective, initially technically successful (as described by the ESVS guidelines11), infrarenal EVAR for unruptured infrarenal AAA;
* Implanted endograft is a Gore Excluder, Medtronic Endurant, Cook Zenith, Cordis Incraft, Endologix AFX, Jotec E-Tegra, or Vascutek Anaconda endograft;
* Follow-up of the AAA of at least one year with imaging of the same modality as the preoperative imaging;
* Axial reconstructions of preoperative CT angiography available, preferably in the arterial phase and with 3 mm or smaller slice thickness.

Exclusion Criteria:

* Patients with ruptured or symptomatic AAA;
* Patients that were treated with fenestrated or branched endografts, iliac branched devices, non-CE marked devices within trial setting, other endografts (EVAS cases) or chimney procedures;
* Acute procedures;
* Reintervention before one year follow-up;
* Revision cases after previous open or endovascular aneurysm repair of an AAA;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, electively treated with EVAR for an infrarenal AAA, will be included from the hospital records of 5 experienced vascular centers, 4 sites in the Netherlands and 1 site in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Prediction model for AAA shrinkage | Preoperative, peroperative and postoperative (until 1-year visit) data
  A prediction model to predict AAA shrinkage one-year after EVAR, it can consist of multiple CTA-scans and/or clinical data.

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (4):
  - Rijnstate Hospital, Arnhem, Non US/Canada
  - Amsterdam UMC, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
- Karolinksa Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] van Rijswijk RE, Bogdanovic M, Roy J, Yeung KK, Zeebregts CJ, Geelkerken RH, Groot Jebbink E, Wolterink JM, Reijnen MMPJ. Multimodal Artificial Intelligence Model for Prediction of Abdominal Aortic Aneurysm Shrinkage After Endovascular Repair ( the ART in EVAR study). J Endovasc Ther. 2025 Jan 30:15266028251314359. doi: 10.1177/15266028251314359. Online ahead of print. PMID 39882767